CLINICAL TRIAL: NCT02632149
Title: The Clinical Research on PINS Vagus Nerve Stimulator for Treatment of Lennox-Gastaut in Children
Brief Title: Trial to Assess Vagus Nerve Stimulation Therapy in Children With Lennox-Gastaut Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Qilu Hospital of Shandong University (Other); Qingdao University (Other); Linyi People's Hospital (Other); Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PINS-017
Record Dates: First submitted 2015-12-13; First posted 2015-12-16 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: PINS Vagus Nerve Stimulator
MeSH Terms: conditions — Lennox Gastaut Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vagus nerve Stimulation is on (Experimental)
  Interventions: Device: PINS Vagus Nerve Stimulator

INTERVENTIONS:
Device: PINS Vagus Nerve Stimulator

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of PINS vagus nerve stimulatior in children with Lennox-Gastaut Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-14 year
2. Lennox - Gastaut syndrome diagnostic standard
3. Regular drug treatment is invalid
4. Antiepileptic drug stability in recent 3 months
5. Good health except epilepsy
6. Patients or his(her) familyscould understand this method and sign the informed consent
7. Patients with good compliance and could complete postoperative follow-up.

Exclusion Criteria:

1. Results of MRI remind epilepsy caused by intracranial space-occupying lesions
2. Had epileptic foci excision surgery or corpus callosum
3. The vagus nerve lesion and damage
4. Tumor, cardiopulmonary anomaly, progressive neurological diseases, asthma， mental disease，peptic ulcer，diabetes Type 1，bad health etc, and other surgical contraindication
5. Participated in other clinical drug test subjects within three months
6. The researchers think that is not suitable for participants'

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluation period 6 month | 6 month of stimulation

SECONDARY OUTCOMES:
Changes in seizure frequency from baseline to the seizure count evaluation period | 1,3,6,months of stimulation
Change from Baseline in the Engel and McHugh description | At 1,3,6 months
Overall WISC Score in Patients from Baseline | Mean change from baseline WISC Overall Score at 1,3,6months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - JiNing First People's Hospital, Jining, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong